CLINICAL TRIAL: NCT04006366
Title: Time Restricted Eating Pilot - Bariatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kelly Allison, Director, Center for Weight and Eating Disorders, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 833432
Record Dates: First submitted 2019-06-26; First posted 2019-07-05 (Actual); Results first posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Time Restricted Feeding
Keywords: bariatrics
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Non-controlled, single arm intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): To test the effects of a 10-hour time restricted eating intervention before and after the 12 weeks of treatment on weight (primary), caloric and macronutrient intake, and a variety of psychosocial measures, including sleep, physical activity, blood pressure and eating behaviors (all secondary).
  Interventions: Behavioral: Time restricted feeding

INTERVENTIONS:
Behavioral: Time restricted feeding — We propose a pilot and feasibility trial of a 10 hour time restricted eating intervention among post-bariatric surgery patients.

SUMMARY:
Bariatric surgery patients have a variable course of weight loss, maintenance and regain. Time restricted eating is an approach that may help individuals lose weight and improve metabolic functioning. We propose a pilot 12-week trial of a 10-hour time restricted eating intervention among post-bariatric surgery patients. The intervention would consist of weekly sessions for 4 weeks, followed by one session every two weeks through 12 weeks, with weight change as the primary outcome.

DETAILED DESCRIPTION:
We propose a pilot 12-week trial of a 10-hour time restricted eating intervention among post-bariatric surgery patients. The intervention would consist of weekly sessions for 4 weeks, followed by one session every two weeks through 12 weeks, with weight change as the primary outcome. We will provide behavioral weight loss education to the patients and monitor how many calories they are taking in once per week.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be at least two years post bariatric surgery who have completed participation in an ongoing longitudinal assessment study of bariatric patients at our medical center.

Exclusion Criteria:

* Participants who were non-compliant with the previous assessment trial, as well as those who were diagnosed with an eating disorder at their final (2 year) assessment visit. We will exclude participants at the discretion of the investigators who have unstable psychiatric issues or would be too ill to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly C Allison, PhD, Principal Investigator — University of Pennyslvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
body mass index [Mean (Standard Deviation); unit: kg/m2] | 40.8 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Compare changes in body weight over 12 weeks in 10 bariatric patients who have undergone bariatric surgery and have completed the pilot study.
Time Frame: baseline to 12 weeks
Population: Six participants enrolled, and 5 completed the trial. We included 5 participants who had more than one data point to calculate weight change.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intervention
Number analyzed (Participants) | 5
kg | -.07 (1.53)

2. Secondary Outcome: Systolic Blood Pressure
Description: Compare changes from baseline to the end of the 12-week intervention in systolic blood pressure.
Time Frame: baseline to 12 weeks
Population: Six participants started the intervention, and we analyzed data from 5 participant who provided blood pressure measurements before and after the intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention
Number analyzed (Participants) | 5
mmHg | 5.4 (14.75)

3. Secondary Outcome: Diastolic Blood Pressure
Description: Compare changes from baseline to the end of the 12-week intervention in diastolic blood pressure.
Time Frame: baseline to 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention
Number analyzed (Participants) | 5
mmHg | -1.8 (6.34)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
This was a small, unfunded feasibility study of this protocol. There was no control group, and no statistical tests were run to test significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT04006366/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT04006366/ICF_001.pdf